CLINICAL TRIAL: NCT01365806
Title: Home ECG Monitoring to Detect Allograft Rejection Following Heart Transplantation
Brief Title: Home Electrocardiogram (ECG) Monitoring After Heart Transplantation
Acronym: NEW HEART
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Francisco (Other); Cedars-Sinai Medical Center (Other); Columbia University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Belinda Chen, Project Director, University of California, Los Angeles
Other Study IDs: 1R01NR012003-01A1 (NIH); 1R01NR012003-01A1 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Transplant Rejection; Qt Interval, Variation in
Keywords: heart transplantation; allograft rejection; QT interval; electrocardiogram (ECG)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The long-term goal of this research is to apply novel technology for detection of donor organ (allograft) rejection to improve patient outcomes following heart transplantation. The specific goal of this study is to determine whether daily monitoring of the transplant recipient's electrocardiogram (ECG) using a simple home device with transmission to an ECG Core Laboratory would provide an early biomarker for acute rejection. Despite routine immunosuppressant drug therapy, acute rejection is common, especially within the first 6 months following transplant surgery. To detect rejection, frequent endomyocardial biopsies of heart tissue are performed. An endomyocardial biopsy is a costly and invasive procedure performed in a hospital cardiac catheterization laboratory that has associated risks. Recent evidence suggests that acute allograft rejection causes delays in ventricular repolarization resulting in a longer QT interval on the ECG. The specific aims of the study are to: 1) determine whether an increase in the QT interval during the first 6 months following heart transplant is a sensitive and specific biomarker for acute rejection; and 2) determine the timing of QT interval increases relative to biopsy-diagnosed stages of mild/moderate/severe rejection. The potential benefit of finding a simple ECG biomarker of allograph rejection that could be measured at home is that it might yield earlier detection of rejection, allow more timely therapy and reduce mortality from acute allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* first heart transplant surgery
* not enrolled in other research studies that conflict with study design

Exclusion Criteria:

* clinically unstable at time of enrollment (i.e. clinical symptoms of allograph impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult heart transplant recipients from recruitment sites (Columbia University-New York Presbyterian Medical Center; University of California, Los Angeles; and Cedars-Sinai Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2011-08; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
number and grade of acute allograft rejection episodes | within one year after transplant surgery

SECONDARY OUTCOMES:
all cause mortality | one year after transplant surgery

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Drew, RN, PhD, FAAN, FAHA, Principal Investigator — University of California, San Francisco; Lynn Doering, RN, DNSc, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - New York Presbyterian-Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Doering LV, Hickey K, Pickham D, Chen B, Drew BJ. Remote noninvasive allograft rejection monitoring for heart transplant recipients: study protocol for the novel evaluation with home electrocardiogram and remote transmission (NEW HEART) study. BMC Cardiovasc Disord. 2012 Mar 2;12:14. doi: 10.1186/1471-2261-12-14. PMID 22386040